CLINICAL TRIAL: NCT02633956
Title: A Phase 2, Randomized, Double Blind, Placebo Controlled Clinical Study Investigating the Effects of Obeticholic Acid and Atorvastatin Treatment on Lipoprotein Metabolism in Subjects With Nonalcoholic Steatohepatitis
Brief Title: Combination Obeticholic Acid (OCA) and Statins for Monitoring of Lipids (CONTROL)
Acronym: CONTROL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intercept Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 747-209
Record Dates: First submitted 2015-11-18; First posted 2015-12-17 (Estimated); Results first posted 2018-06-04 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Nonalcoholic Steatohepatitis
Keywords: Non-alcoholic Fatty Liver Disease; NAFLD; Fatty Liver Disease; NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — obeticholic acid; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 5 mg Obeticholic Acid (Experimental): 5 mg Obeticholic Acid daily for the double-blind treatment period. 10 mg Atorvastatin titrating to 20mg.
  Interventions: Drug: Obeticholic Acid; Drug: Atorvastatin
- 10 mg Obeticholic Acid (Experimental): 10 mg Obeticholic Acid daily for the double-blind treatment period. 10 mg Atorvastatin titrating to 20mg.
  Interventions: Drug: Obeticholic Acid; Drug: Atorvastatin
- 25 mg Obeticholic Acid (Experimental): 25 mg Obeticholic Acid daily for the double-blind treatment period. 10 mg Atorvastatin titrating to 20mg.
  Interventions: Drug: Obeticholic Acid; Drug: Atorvastatin
- Placebo (Placebo Comparator): One tablet daily for the double-blind treatment period. 10 mg Atorvastatin titrating to 20mg.
  Interventions: Drug: Atorvastatin; Drug: Placebo

INTERVENTIONS:
Drug: Obeticholic Acid — Once a day (QD) by mouth (PO)
  Other Names: OCA; 6alpha-ethylchenodeoxycholic acid (6-ECDCA); INT-747
  Arms: 10 mg Obeticholic Acid; 25 mg Obeticholic Acid; 5 mg Obeticholic Acid
Drug: Atorvastatin — Initiate treatment with Atorvastatin at Week 4 visit with a dose of 10 mg once daily (QD) by mouth (PO).
  Increase Atorvastatin to 20 mg once daily (QD) by mouth (PO) at Week 8 visit if 10 mg daily is tolerated.
  Atorvastatin may be titrated up or down at Week 12 visit as clinically indicated.
Drug: Placebo — Once a day (QD) by mouth (PO)
  Arms: Placebo

SUMMARY:
This Phase 2, double-blind, randomized, placebo-controlled, multicenter study, with an open-label long-term safety extension (LTSE), will evaluate the effect of Obeticholic Acid, and the subsequent addition of statin therapy, on lipoprotein metabolism in subjects with nonalcoholic steatohepatitis (NASH) with fibrosis stage 1 to 4, but no evidence of hepatic decompensation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Histologic evidence of NASH, as assessed by central reading of a liver biopsy obtained no more than 1 year prior to randomization, defined by the presence of all 3 key histological features of NASH with a score of at least 1 for each and a combined score of 4 or greater out of a possible 8 points according to NASH Clinical Research Network (CRN) criteria.
3. Histologic evidence of fibrosis stage 1 to stage 4 (as defined by NASH CRN scoring of fibrosis) without any evidence of hepatic decompensation.
4. If subject has type 2 diabetes, is on stable dose of anti-diabetic medication (except thiazolidinediones [TZDs]) for ≥3 months prior to Day 1.
5. Is either not taking or is on stable doses of TZDs and/or Vitamin E for ≥6 months prior to Day 1.
6. Contraception: Female subjects of childbearing potential must use ≥1 effective method of contraception during the study and until 30 days following the last dose of investigational product. Effective methods of contraception are considered to be the following: barrier method, ie, condom (male or female) with spermicide or diaphragm with spermicide, intrauterine device, vasectomy (partner), hormonal (eg, contraceptive pill, patch, intramuscular implant or injection), abstinence (defined as refraining from heterosexual intercourse).
7. Must provide written informed consent and agree to comply with the study protocol, including adherence to protocol-described statin withdrawal and statin therapy.

Exclusion Criteria:

1. Current or history of significant alcohol consumption for a period of more than 3 consecutive months within 1 year prior to Screening Visit 1 (significant alcohol consumption is defined as more than 2 units/day in females and more than 4 units/day in males, on average)
2. Prior intolerance to treatment with atorvastatin or other 3-hydroxy-3-methyl-glutaryl (HMG) Coenzyme A reductase inhibitors (including but not limited to rhabdomyolysis).
3. LDL cholesterol ≥190 mg/dL and already on statin therapy at Screening Visit 1.
4. LDL cholesterol >200 mg/dL at any Screening Visit in subjects who are not on statin therapy, or at Screening Visit 2 in statin washout subjects.
5. Planned change in diet or exercise habits during participation in the double-blind period, or a significant weight change of >5% in the prior 6 months.
6. Subjects who have undergone gastric bypass procedures (gastric lap band is acceptable) or ileal resection or plan to undergo either of these procedures.
7. History of biliary diversion
8. Uncontrolled diabetes defined as HbA1c ≥9.5% within 60 days prior to randomization (Day 1).
9. Administration of any of the following medications as specified below:

   * Prohibited 30 days prior to Day 1:

     * bile acid sequestrants (BAS) including cholestyramine and its derivatives, colesevelam, colestipol, or
     * omega-3 fatty acid-containing dietary supplements
   * Prohibited 3 months prior to Day 1:

     * nicotinic acid and derivatives, ezetimibe
     * any prescription or over-the-counter (OTC) medication or herbal remedy with putative NASH efficacy (except Vitamin E or TZDs)
     * ursodeoxycholic acid
     * fenofibrate or other fibrates
     * any OTC or health food used to treat lipids including plant sterols and berberine
   * Prohibited 6 months prior to Day 1:

     * azathioprine, colchicine, cyclosporine, methotrexate, mycophenolate, mofetil, pentoxifylline; budesonide and other systemic corticosteroids, or
     * potentially hepatotoxic drugs (including α-methyl-dopa, sodium valproic acid, isoniazide, or nitrofurantoin)
   * Prohibited 12 months prior to Day 1:

     * antibodies or immunotherapy directed against interleukins, or
     * other cytokines or chemokines
10. Evidence of other forms of chronic liver disease including but not limited to:

    * Positive test result at Screening for hepatitis B surface antigen
    * Active hepatitis C virus (HCV) infection (positive for HCV ribonucleic acid [RNA] at Screening) or history of positive HCV RNA test result
    * Primary biliary cirrhosis, primary sclerosing cholangitis, autoimmune hepatitis or overlap syndrome
    * Alcoholic liver disease
    * Wilson's disease or hemochromatosis or iron overload
    * Alpha-1-antitrypsin (A1AT) deficiency
    * Prior known drug-induced liver injury within 5 years before Day 1
    * Known or suspected hepatocellular carcinoma
11. History of liver transplant, current placement on a liver transplant list, or current Model for End-Stage Liver Disease (MELD) score >12. Subjects who are placed on a transplant list despite relatively early disease stage (eg, per regional guidelines) may be eligible as long as they do not meet any of the other exclusion criteria
12. Presence of hepatic decompensation, including:

    * Gastroesophageal varices
    * Ascites
    * Hepatic encephalopathy
    * Spontaneous bacterial peritonitis
    * Hepatorenal or hepatopulmonary syndromes
13. Total bilirubin ≥2x upper limit of normal (ULN) at any Screening Visit (subjects with Gilbert's syndrome may be enrolled despite a total bilirubin level >2x ULN if their conjugated bilirubin is <2x ULN)
14. Creatine phosphokinase >5x ULN at Screening Visit 2
15. Serum creatinine ≥1.5 mg/dL at any Screening Visit
16. Serum alanine aminotransferase (ALT) >300 U/L at any Screening Visit
17. Platelet count <75,000/mm3 at any Screening Visit
18. Known positivity for human immunodeficiency virus (HIV) infection
19. Subjects with recent history (within 1 year of randomization) of cardiovascular disease or with history or planned cardiovascular interventions to treat atherosclerotic cardiovascular disease
20. Other concomitant disease, malignancy, or condition likely to significantly decrease life expectancy to <5 years, including known cancers (except carcinomas in situ or other stable, relatively benign conditions such as chronic lymphocytic leukemia) and moderate to severe congestive heart failure.
21. Known substance abuse, including inhaled or injected drugs in the year before Screening.
22. For female subjects: pregnancy, planned or potential for pregnancy and unwillingness to use effective birth control during the study, or breastfeeding
23. Participation in a clinical research study with any investigational product being evaluated for the treatment of diabetes or NASH in the 6 months before Day 1.
24. Receipt of any investigational product not being evaluated for the treatment of diabetes or NASH from Screening Visit 1 to Day 1, within 30 days prior to Day 1, or within 5 half-lives of the compound before Day 1 (whichever was longer)
25. Previous exposure to Obeticholic Acid
26. History of known or suspected clinically significant hypersensitivity to Obeticholic Acid or any of its components
27. Mental instability or incompetence, such that the validity of informed consent or ability to be compliant with the study is uncertain
28. Any other condition which, in the opinion of the Investigator, would impede compliance or hinder completion of the study
29. Acute cholecystitis or acute biliary obstruction

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-12-04 (Actual); Primary Completion 2017-03-21 (Actual); Study Completion 2018-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Shapiro, MD, Study Director — Intercept Pharmaceuticals
Locations (22):
- United States (22):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Scripps Clinic, La Jolla, California
  - Inland Empire Liver Foundation, Rialto, California
  - Nature Coast Clinical Research, Inverness, Florida
  - University of Miamai, Schiff Center for Liver Diseases, Miami, Florida
  - South Florida Center of Gastroenterology, Wellington, Florida
  - Florida Medical Clinic, P.A., Zephyrhills, Florida
  - The Queen's Medical Center - Liver Center, Honolulu, Hawaii
  - Mercy Medical Center, Institute for Digestive Health & Liver Disease, Baltimore, Maryland
  - Kansas City Research Institute, Kansas City, Missouri
  - St. Louis University, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University Gastroenterology Liver Center, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - ClinSearch, Chattanooga, Tennessee
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - Liver Associates of Texas, P.A., Houston, Texas
  - American Research Corporation at the Texas Liver Institute, San Antonio, Texas
  - McGuire DVAMC, Richmond, Virginia

REFERENCES:
- [Derived] Pockros PJ, Fuchs M, Freilich B, Schiff E, Kohli A, Lawitz EJ, Hellstern PA, Owens-Grillo J, Van Biene C, Shringarpure R, MacConell L, Shapiro D, Cohen DE. CONTROL: A randomized phase 2 study of obeticholic acid and atorvastatin on lipoproteins in nonalcoholic steatohepatitis patients. Liver Int. 2019 Nov;39(11):2082-2093. doi: 10.1111/liv.14209. Epub 2019 Sep 10. PMID 31402538

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects using statins within 30 days of the initial Screening visit (Screening Visit 1) are required to stop statin therapy immediately following this initial visit and must undergo a 4-week statin washout period prior to Screening Visit 2.
Groups:
- 5 mg Obeticholic Acid: 5 mg Obeticholic Acid daily for the double-blind treatment period. 10 mg Atorvastatin titrating to 20mg.
  Obeticholic Acid: Once a day (QD) by mouth (PO)
  Atorvastatin: Initiate treatment with Atorvastatin at Week 4 visit with a dose of 10 mg once daily (QD) by mouth (PO).
  Increase Atorvastatin to 20 mg once daily (QD) by mouth (PO) at Week 8 visit if 10 mg daily is tolerated.
  Atorvastatin may be titrated up or down at Week 12 visit as clinically indicated.
- 10 mg Obeticholic Acid: 10 mg Obeticholic Acid daily for the double-blind treatment period. 10 mg Atorvastatin titrating to 20mg.
  Obeticholic Acid: Once a day (QD) by mouth (PO)
  Atorvastatin: Initiate treatment with Atorvastatin at Week 4 visit with a dose of 10 mg once daily (QD) by mouth (PO).
  Increase Atorvastatin to 20 mg once daily (QD) by mouth (PO) at Week 8 visit if 10 mg daily is tolerated.
  Atorvastatin may be titrated up or down at Week 12 visit as clinically indicated.
- 25 mg Obeticholic Acid: 25 mg Obeticholic Acid daily for the double-blind treatment period. 10 mg Atorvastatin titrating to 20mg.
  Obeticholic Acid: Once a day (QD) by mouth (PO)
  Atorvastatin: Initiate treatment with Atorvastatin at Week 4 visit with a dose of 10 mg once daily (QD) by mouth (PO).
  Increase Atorvastatin to 20 mg once daily (QD) by mouth (PO) at Week 8 visit if 10 mg daily is tolerated.
  Atorvastatin may be titrated up or down at Week 12 visit as clinically indicated.
- Placebo: One tablet daily for the double-blind treatment period. 10 mg Atorvastatin titrating to 20mg.
  Atorvastatin: Initiate treatment with Atorvastatin at Week 4 visit with a dose of 10 mg once daily (QD) by mouth (PO).
  Increase Atorvastatin to 20 mg once daily (QD) by mouth (PO) at Week 8 visit if 10 mg daily is tolerated.
  Atorvastatin may be titrated up or down at Week 12 visit as clinically indicated.
  Placebo: Once a day (QD) by mouth (PO)
Period: Overall Study
Arm/Group | 5 mg Obeticholic Acid | 10 mg Obeticholic Acid | 25 mg Obeticholic Acid | Placebo
Started | 20 | 21 | 22 | 21
Completed | 19 | 19 | 20 | 21
Not Completed | 1 | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5 mg Obeticholic Acid | 10 mg Obeticholic Acid | 25 mg Obeticholic Acid | Placebo | Total
Number analyzed (Participants) | 20 | 21 | 22 | 21 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (10.13) | 57.1 (11.62) | 62.2 (11.06) | 59.8 (9.88) | 58.1 (11.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 10 | 13 | 51
  Male | 4 | 9 | 12 | 8 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 5 | 4 | 20
  Not Hispanic or Latino | 13 | 17 | 17 | 17 | 64
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 1 | 0 | 2 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1 | 2
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 19 | 20 | 19 | 16 | 74
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Fibrosis stage (NASH Clinical Research Network (CRN) categories) [Count of Participants; unit: Participants] — The NASH CRN Fibrosis Staging is based on the degree of liver fibrosis from Stage 0: no fibrosis to Stage 4: cirrhosis. The related histological classification of each stage is as follows: Fibrosis Stage: Stage 0: none; Stage 1a: zone 3 perisinusoidal, delicate; 1b: zone 3 perisinusoidal, dense; 1c: portal only; Stage 2: 1a or 1b + periportal fibrosis; Stage 3: bridging fibrosis; and Stage 4: cirrhosis.
  The higher the fibrosis stage the worse the prognosis.
  Participants
    Stage 1 and 2 | 10 | 10 | 11 | 10 | 41
    Stage 3 and 4 | 10 | 11 | 11 | 11 | 43
Screening LDL [Count of Participants; unit: Participants] — Fasting LDL concentration
  Participants
    Less than or equal 125 mg/dL | 11 | 11 | 13 | 11 | 46
    Greater than 125 mg/dL | 9 | 10 | 9 | 10 | 38

OUTCOME MEASURES:

1. Primary Outcome: The Effect of Obeticholic Acid on Low-density Lipoprotein (LDL) Concentration (Least Squares Mean Change From Baseline at Week 16)
Description: The effect of Obeticholic Acid on LDL metabolism in subjects with biopsy confirmed nonalcoholic steatohepatitis (NASH) and the ability of atorvastatin to modulate this effect as measured by change (least squares mean) from baseline at week 16 in LDL concentration
Time Frame: Baseline and Week 16
Population: Efficacy evaluable population
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | 5 mg Obeticholic Acid | 10 mg Obeticholic Acid | 25 mg Obeticholic Acid | Placebo
Number analyzed (Participants) | 13 | 17 | 18 | 19
mg/dL | -33.2 (4.93) | -44.27 (4.10) | -39.54 (4.24) | -53.33 (3.93)
Statistical Analysis 1: Comparison: 25 mg Obeticholic Acid vs Placebo; Test type: Other — Estimation; Least Square Mean Difference = 13.79, 95% CI 2-sided [2.28 to 25.30], Standard Error of Mean 5.75
Statistical Analysis 2: Comparison: 10 mg Obeticholic Acid vs Placebo; Test type: Other — Estimation; Least Square Mean Difference = 9.06, 95% CI 2-sided [-2.18 to 20.30], Standard Error of Mean 5.61
Statistical Analysis 3: Comparison: 5 mg Obeticholic Acid vs Placebo; Test type: Other — Estimation; Least Square Mean Difference = 20.13, 95% CI 2-sided [7.33 to 32.92], Standard Error of Mean 6.39

2. Primary Outcome: The Effect of Obeticholic Acid on LDL Particle Size (Least Squares Mean Change From Baseline at Week 16)
Description: The effect of Obeticholic Acid on LDL metabolism in subjects with biopsy confirmed NASH and the ability of atorvastatin to modulate this effect as measured by change from baseline (least squares mean) at week 16 in LDL particle size. It is LDL particle diameter size (nm) that is reported.
Time Frame: Baseline and Week 16
Population: Efficacy evaluable population
Measure: Least Squares Mean (Standard Error); unit: nm
Arm/Group | 5 mg Obeticholic Acid | 10 mg Obeticholic Acid | 25 mg Obeticholic Acid | Placebo
Number analyzed (Participants) | 12 | 17 | 17 | 17
nm | 0.02 (0.15) | -0.41 (0.12) | -0.09 (0.12) | -0.49 (0.12)
Statistical Analysis 1: Comparison: 25 mg Obeticholic Acid vs Placebo; Test type: Other — Estimation; Least Square Mean Difference = 0.41, 95% CI 2-sided [0.07 to 0.75], Standard Error of Mean 0.17
Statistical Analysis 2: Comparison: 10 mg Obeticholic Acid vs Placebo; Test type: Other — Estimation; Least Square Mean Difference = 0.09, 95% CI 2-sided [-0.25 to 0.42], Standard Error of Mean 0.17
Statistical Analysis 3: Comparison: 5 mg Obeticholic Acid vs Placebo; Test type: Other — Estimation; Least Square Mean Difference = 0.51, 95% CI 2-sided [0.14 to 0.89], Standard Error of Mean 0.19

3. Primary Outcome: The Effect of Obeticholic Acid on LDL Particle Concentration (Total) (Least Squares Mean Change From Baseline at Week 16)
Description: The effect of Obeticholic Acid on LDL metabolism in subjects with biopsy confirmed nonalcoholic NASH and the ability of atorvastatin to modulate this effect as measured by change (least squares mean) from baseline at week 16 in LDL particle concentration (total)
Time Frame: Baseline and Week 16
Population: Efficacy evaluable population
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | 5 mg Obeticholic Acid | 10 mg Obeticholic Acid | 25 mg Obeticholic Acid | Placebo
Number analyzed (Participants) | 12 | 17 | 17 | 19
nmol/L | -224.79 (62.58) | -325.04 (49.81) | -336.22 (51.40) | -439.84 (47.70)
Statistical Analysis 1: Comparison: 25 mg Obeticholic Acid vs Placebo; Test type: Other — Estimation; Least Square Mean Difference = 103.61, 95% CI 2-sided [-35.58 to 242.81], Standard Error of Mean 69.51
Statistical Analysis 2: Comparison: 10 mg Obeticholic Acid vs Placebo; Test type: Other — Estimation; Least Square Mean Difference = 114.80, 95% CI 2-sided [-21.53 to 251.13], Standard Error of Mean 68.08
Statistical Analysis 3: Comparison: 5 mg Obeticholic Acid vs Placebo; Test type: Other — Estimation; Least Square Mean Difference = 215.05, 95% CI 2-sided [55.84 to 374.26], Standard Error of Mean 79.51

ADVERSE EVENTS:
Time Frame: From time of first dose to end of double-blind phase participation, up to 16 weeks
Arm/Group | 5 mg Obeticholic Acid | 10 mg Obeticholic Acid | 25 mg Obeticholic Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21 | 0/22 | 0/21
Serious Adverse Events (participants affected / at risk) | 2/20 | 1/21 | 1/22 | 0/21
Other Adverse Events (participants affected / at risk) | 13/20 | 9/21 | 19/22 | 9/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg Obeticholic Acid (N=20) | 10 mg Obeticholic Acid (N=21) | 25 mg Obeticholic Acid (N=22) | Placebo (N=21)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg Obeticholic Acid (N=20) | 10 mg Obeticholic Acid (N=21) | 25 mg Obeticholic Acid (N=22) | Placebo (N=21)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 12 (19) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 0 (0) | 2 (2) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 3 (3) | 3 (3) | 1 (1)
Weight increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators must wait 18 months after the study end to publish their results and a multi-center publication must come first. The sponsor has a 45 day review period with the option to extend to an additional 90 days.

DOCUMENTS (2):
  • Study Protocol (2016-12-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT02633956/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-20): https://cdn.clinicaltrials.gov/large-docs/56/NCT02633956/SAP_001.pdf